CLINICAL TRIAL: NCT00731822
Title: Study HZC111348, a Repeat-dose Study of GW685698/GW642444 Inhalation Powder Versus Placebo in the Treatment of Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study To Assess Single Dosage Strength Of GW685698/GW642444 Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZC111348
Record Dates: First submitted 2008-08-08; First posted 2008-08-11 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; Novel Dry Powder Inhaler; Chronic Obstructive Pulmonary Disease (COPD); GW685698/GW642444
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Drug: GW685698/GW642444 — GW685698/GW642444

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a single dosage strength of GW685698/GW642444 in subjects with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria:

1. Informed consent: Subjects must give their signed written informed consent to participate.
2. Gender: Male subjects or female subjects of non-child bearing potential (e.g. post-menopausal or surgical sterile) 40 - 80 years of age at screening (Visit 1).

   * Post-menopausal females are defined as being amenorrhoeic for greater than 2 years with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. However if indicated this can be confirmed by estradiol and FSH levels consistent with menopause (according to laboratory ranges) at screening (Visit 1).
   * Surgically sterile females are defined as those with a documented (medical report verification) hysterectomy and/or bilateral oophorectomy or Tubal Ligation.
   * Furthermore, male subjects in this study must use double-barrier (condom/spermicide) birth control methods or abstain from sexual intercourse with female partners who are pregnant, lactating, or able to bear children in addition to any birth control methods the female partner is using, from the first dose of the study medication until 90 days after the last dose of the study medication.
3. COPD diagnosis: Subjects with a clinical history of COPD in accordance with the following definition by the American Thoracic Society/European Respiratory Society [Celli, 2004] :

   COPD is a preventable and treatable disease characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.
4. Tobacco use: subjects with a current or previous history of ≥ 10 pack-years of cigarette smoking at screening (Visit 1). Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.

   • Number of pack years = (number of cigarette per day/20)) x number of years smoked
5. Severity of Disease: subjects who conform to the current severity classification for Stage II/III disease in terms of post-bronchodilator spirometry at Screening Visit 1:

   * Subject with a measured post-salbutamol FEV1/FVC ratio of ≤0.70
   * Subjects with a measured post-salbutamol FEV1 ≥ 40 % and ≤ 80 % of predicted normal values calculated using NHANES III reference equations.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Pregnancy: Women who are pregnant or lactating
2. Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if COPD is the current diagnosis)
3. α1- antitrypsin deficiency: Subjects with α-1 antitrypsin deficiency as the underlying cause of COPD
4. Other respiratory disorders: Subjects with active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
5. Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening
6. Chest X-ray (or CT scan): Subjects with a chest X-ray (or CT scan) that reveals evidence of clinically significant abnormalities not believed to be due to the presence of COPD. A chest X-ray must be taken at Screening if a chest X-ray or CT scan is not available within 6 months prior to Screening
7. Poorly controlled COPD: Subjects with poorly controlled COPD, defined as the occurrence of any of the following in the 6 weeks prior to Screening:

   * Acute worsening of COPD that is managed by subject with corticosteroids or antibiotics, or
   * Acute worsening of COPD that requires treatment prescribed by a physician Subjects who are hospitalized due to poorly controlled COPD within 12 weeks of the Screening Visit
8. Lower respiratory tract infection: Subjects with lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to Visit 1
9. 12-lead ECG (Electrocardiogram): An abnormal and clinically significant 12-lead ECG that results in an active medical problem. For this study, an abnormal ECG is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following:

   * Clinically significant conduction abnormalities (e.g. left bundle branch block, Wolff-Parkinson-White syndrome)
   * Clinically significant arrhythmias (e.g. atrial fibrillation, ventricular tachycardia)

   The independent cardiologist, contracted by GSK, will determine the clinical significance of any ECG abnormalities and determine if a subject is precluded from entering the study. However, the following predetermined ECG abnormalities are considered clinically significant and will result in exclusion of a subject:
   * Ventricular rate < 45 bpm
   * PR interval > 240 msec
   * Evidence of Second-Degree (Mobitz type II) or Third-Degree atrioventricular (AV) block
   * Pathological Q waves
   * Non-specific intraventricular conduction delay
   * ST-T wave abnormalities (excluding non-specific ST-T wave abnormalities)
   * Right or left complete bundle branch block
   * A mean QTc(B) value at Screening > 450 msec, or uncorrected QT >600 msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T wave)
10. Other Diseases/abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
11. Hepatitis: Subjects with a positive Hepatitis B surface antigen or positive Hepatitis C antibody pre-study or at Screening
12. Hypertension: Subjects with clinically significant hypertension that is uncontrolled
13. Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years.

    • Carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded if the subject has been considered cured within 5 years since diagnosis.
14. Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medications (e.g. beta-agonists, corticosteroid) or components of the inhalation powder (e.g. lactose, magnesium stearate). Or a history of drug or other allergy such as a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates the subject's participation
15. Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years
16. Medication prior to spirometry: Subjects who are medically unable to withhold their rescue medication for the 6-hour period required prior to spirometry testing at each study visit.
17. Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen prn use (i.e. ≤ 12 hours per day) is not exclusionary.
18. Pulmonary rehabilitation: Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Programme within 4 weeks prior to Screening or who will enter the acute phase of a Pulmonary Rehabilitation Programme during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Programme may be included.
19. Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures
20. Questionable validity of Consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study
21. Prior use of study medication/other investigational drugs: Subjects who have received the GW642444 in previous studies. Subjects who have received an investigational drug within 30 days of entry into this study (Screening), or within 5 drug half-lives of the investigational drug, whichever is longer
22. Sleep apnea: Subjects with clinically significant sleep apnea that is uncontrolled.
23. Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Norway (5):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Sandvika
  - GSK Investigational Site, Trondheim
- Sweden (4):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Luleå
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Lotvall J, Bakke PS, Bjermer L, Steinshamn S, Scott-Wilson C, Crim C, Sanford L, Haumann B. Efficacy and safety of 4 weeks' treatment with combined fluticasone furoate/vilanterol in a single inhaler given once daily in COPD: a placebo-controlled randomised trial. BMJ Open. 2012 Jan 19;2(1):e000370. doi: 10.1136/bmjopen-2011-000370. Print 2012. PMID 22267687
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: HZC111348 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HZC111348 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HZC111348 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HZC111348 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HZC111348 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HZC111348 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HZC111348 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting eligibility criteria at screening and randomization criteria at the end of the Screening Period (SP) were randomized to 1 of 2 treatments: Fluticasone Furoate (FF)/Vilanterol (GW642444) 400/25 microgram (µg) inhalation powder or matching placebo. 89 participants were screened, of whom 60 were randomized.
Groups:
- Placebo: Participants received matching placebo once daily (OD) in the morning via a dry powder inhaler (DPI) for 28 days.
- FF/VI 400/25 µg OD: Participants received fluticasone furoate (FF)/Vilanterol (VI [GW642444]) 400/25 micrograms (µg) OD in the morning via a DPI for 28 days.
Period: Overall Study
Arm/Group | Placebo | FF/VI 400/25 µg OD
Started | 20 | 40
Completed | 16 | 39
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF/VI 400/25 µg OD | Total
Number analyzed (Participants) | 20 | 40 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (6.01) | 63.5 (7.10) | 63.6 (6.71)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 15 | 20
  Male | 15 | 25 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 40 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted Mean Heart Rate 0-4 Hours Post-dose at the End of the 28-day Treatment Period
Description: Co-Primary Endpoint. Weighted mean was derived by calculating the average area under the curve (AUC), and then dividing by the relevant time interval. Baseline is the most recent result taken on or before pre-dose Day 1. Heart rate was recorded at 60 minutes (min) prior to dosing and at 15 min, 45 min, 90 min, 120 min, and 240 min post-dose on Day 28. Change from Baseline was calculated as the Day 28 value minus the Baseline value. Analysis was performed using a restricted maximum likelihood (REML)-based repeated measures mixed model approach (MMRM) with covariates of Baseline heart rate, sex, age, smoking status, treatment, and day and day by treatment and day by Baseline interactions. par.=participants.
Time Frame: Baseline to Day 28
Population: Intent-to-Treat (ITT) Population: all randomized par. who received at least one dose of study medication. The number of par. presented represent those with data available at the time point being presented; however, all par. in the ITT Population without missing covariate information and with >=1 post-BL measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute (bpm)
Arm/Group | Placebo | FF/VI 400/25 µg OD
Number analyzed (Participants) | 20 | 40
Beats per minute (bpm) | -5.7 (1.83) | -5.1 (1.23)
Statistical Analysis 1: Comparison: Placebo vs FF/VI 400/25 µg OD; Test type: Superiority or Other; Least Squares Mean Difference = 0.6, 95% CI 2-sided [-3.9 to 5.1]

2. Primary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE) Throughout the Study
Description: Co-Primary Endpoint. An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; or is a congenital anomaly/birth defect. See the SAE/AE module of this results summary for a list of specific SAEs/AEs occurring in the study.
Time Frame: From Baseline (Day 1) until Follow-up (up to Study Day 37)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | FF/VI 400/25 µg OD
Number analyzed (Participants) | 20 | 40
participants
  Any AE | 10 | 27
  Any SAE | 0 | 1

3. Secondary Outcome: Mean Change From Baseline in Clinic Visit Trough Forced Expiratory Volume in One Second (FEV1) on Days 2, 15, and 29
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Days 2, 15, and 29 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Days 1, 14, and 28. The highest of 3 technically acceptable measurements was recorded. Baseline FEV1 is defined as the mean of the two assessments obtained 30 minutes pre-dose and immediately pre-dose on Day 1. Change from Baseline was calculated as the Day 29 value minus the Baseline value. Analysis was performed using Mixed Model Repeated Measures (MMRM) with covariates of Baseline FEV1, sex, age, smoking status, treatment and day, and day by treatment and day by Baseline interactions.
Time Frame: Baseline; Day 2, Day 15, and Day 29
Population: ITT Population. The number of participants presented (indicated by n=X, X in the category titles) represents the number of participants with data available at that time point. However all participants in the ITT Population without missing covariate information and with at least one post-Baseline measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF/VI 400/25 µg OD
Number analyzed (Participants) | 20 | 40
Liters
  Day 2, n=20, 39 | 0.122 (0.0323) | 0.276 (0.0229)
  Day 15, n=15, 39 | 0.113 (0.0387) | 0.285 (0.0253)
  Day 29, n=16, 39 | 0.088 (0.0398) | 0.271 (0.0262)

4. Secondary Outcome: Mean Change From Baseline (Pre-dose on Day 1) in Weighted Mean FEV1 (0-4 Hours Post-dose) on Days 1 and 28
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry at the Day 1 and Day 28 clinic visits (60 minutes pre-dose; immediately pre-dose; post-dose after 5, 15, and 30 minutes and 1, 2, and 4 hours. Weighted mean was calculated using the 24-hour serial FEV1 measurements that included the 0 to 4 hours post-dose assessment. At each time point, the highest of 3 technically acceptable measurements was recorded. Baseline FEV1 was defined as the mean of the two assessments obtained 30 minutes pre-dose and immediately pre-dose on Day 1. Change from Baseline was calculated as the average Day 28 FEV1 value minus the Baseline value. Analysis was performed using Mixed Model Repeated Measures (MMRM) with covariates of Baseline FEV1, sex, age, smoking status, treatment and day, and day by treatment and day by Baseline interactions.
Time Frame: Baseline (pre-dose on Day 1); Day 1 and Day 28
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF/VI 400/25 µg OD
Number analyzed (Participants) | 20 | 40
Liters
  Day 1, n=20, 40 | 0.022 (0.0259) | 0.222 (0.0182)
  Day 28, n=16, 39 | 0.047 (0.0341) | 0.283 (0.0227)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication through the study treatment stop date (Day 28 +1).
Description: An on-therapy AE or SAE is defined as an AE with an onset on or after the start date of study medication, but not later than one day after the last date of study medication. SAEs and AEs were collected in members of the ITT Population, comprised of all participants randomized to treatment, who received at least one dose of the study medication.
Arm/Group | Placebo | FF/VI 400/25 µg OD
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/40
Other Adverse Events (participants affected / at risk) | 10/20 | 16/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | FF/VI 400/25 µg OD (N=40)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | FF/VI 400/25 µg OD (N=40)
Nasopharyngitis (Infections and infestations) | 3 | 7
Oral candidiasis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 6
Dizziness (Nervous system disorders) | 1 | 2
Chest pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.